CLINICAL TRIAL: NCT03637075
Title: Characterization of Insulin Action and Dopamine-signaling in the Human Brain of Normal Weight and Obese Subjects by [11C]-Raclopride-PET/MRT
Brief Title: Raclopride-PET/MRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: GK-PET/MR Tü-014
Record Dates: First submitted 2018-08-03; First posted 2018-08-17 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes mellitus, Type 2; cerebral insulin resistance; insulin action in the human brain; dopamine signalling
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: single-blinded, monocentric, prospective crossover study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Intranasal placebo administration
  Interventions: Other: Placebo
- Intranasal insulin (Active Comparator): Intranasal insulin administration
  Interventions: Other: intranasal insulin

INTERVENTIONS:
Other: intranasal insulin — intranasal administration of insulin (160 IU)
  Arms: Intranasal insulin
Other: Placebo — placebo intranasal administration
  Arms: Placebo

SUMMARY:
Cerebral insulin resistance plays an important role in the development of obesity and diabetes mellitus type 2. The aim of this project is to examine the effect of human nasal insulin on the dopaminergic system. Therefore, characteristics of cerebral dopamine receptors before and after administration of nasal insulin vs. placebo shall be analyzed in a randomized way. Moreover, the investigators plan to examine the insulin action on cortical and subcortical activation in humans and the interaction of dopamine metabolism with [11C]-Raclopride-PET/MRI. By performing fMRI measurements, insulin sensitivity of the central nervous system can be investigated simultaneously. Recruiting is planed as a two-step process.First 12 normal-weight (BMI 20-25 kg/m²) men should be examined. If first results show a insulin-dependent effect on the availability of dopamine receptors in the human brain, recruitment of 12 overweight men will get started.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures.
* Intake of any medication
* HbA1C <6%
* BMI 20-25 kg/m²
* Clinical routine blood parameters within the normal ranges
* All participants must agree to get informed of unexpected detected, clinical relevant findings.

Exclusion Criteria:

* Acute diseases such as infections (e.g.)
* Any relevant cardiovascular disease
* Any surgery within the last three months
* Any neurologic or psychiatric disease
* Known allergies
* Hb < 13 g/dl
* Presence of any contraindication for the conduct of an MRI investigation, such as cardiac pacemakers, ferromagnetic haemostatic clips in the central nervous system, metallic splinters in the eye, ferromagnetic or electronically operated active devices like automatic cardioverter defibrillators, cochlear implants, insulin pumps and nerve stimulators, prosthetic heart valves etc.
* Claustrophobia

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Effects of nasal insulin vs. placebo on the insulin sensitivity of the human brain as well as effects on regional availability of dopamine receptors. | 0-60 min
  assessed by fMRI (insulin sensitivity of the brain measured as change in regional brain activity and Raclopride-PET/MRT (regional dopamine receptor availability).

SECONDARY OUTCOMES:
Differences between normalweight and overweight subjects regarding insulin sensitivity and availability of dopamine receptors | 0 - 60 min
  assessed by fMRI and Raclopride-PET/MRT
Effects of nasal insulin vs. placebo on changes in plasma insulin levels | 0 - 60min
  assessed by blood sampling after application.
Effects of nasal insulin vs. placebo on changes in plasma glucose levels | 0 - 60min
  assessed by blood sampling after application.
Effects of nasal insulin vs. placebo on changes in FFA levels | 0 - 60min
  assessed by blood sampling after application.
Effects of nasal insulin vs. placebo on changes in prolactin levels as a proxy for the dopaminergic tonus | 0 - 60min
  assessed by blood sampling after application.
Effects of nasal insulin vs. placebo on changes in autonomic nervous system | -30 - 60 min
  assessed by heart rate variability.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tuebingen, Department of Internal Medicine IV, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No